CLINICAL TRIAL: NCT02956590
Title: Dyslipidemia of Obesity Intervention in Teens Trial
Brief Title: Dyslipidemia of Obesity Intervention in Teens
Acronym: DO IT!
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHN DO IT!
Record Dates: First submitted 2016-10-21; First posted 2016-11-07 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Dyslipidemia; Obesity
Keywords: dyslipidemia; obesity; pitavastatin; lipids
MeSH Terms: conditions — Dyslipidemias; Obesity | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pitavastatin (Active Comparator): Study Drug
  Interventions: Drug: Pitavastatin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitavastatin — Statin
  Other Names: Livalo
  Arms: Pitavastatin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This trial of pitavastatin will determine efficacy and safety in this high risk population and provide evidence for clinicians to target this treatable risk factor to achieve an impact on early atherosclerosis, and potentially achieve primary prevention of adult cardiovascular disease.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled clinical trial of pitavastatin for 2 years comparing the effect of study drug versus placebo on vascular measures in at least 354 adolescents with excess adiposity and CDO (defined as high non-HDL-C + high triglycerides (TG)/HDL-C ratio or low HDL-C). Enrollment will take place over 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls aged 10 to 19 years (with 2-year availability for study participation)
* BMI ≥85th percentile (using Centers for Disease Control (CDC) BMI charts)
* Fasting lipid profile x2 each with all of the following:

  * LDL-C <160 mg/dL and ≥90 mg/dL, and
  * TG (triglycerides) <500 mg/dL, and
  * TG/HDL-C ratio ≥2.5 or HDL-C <45 mg/dL for boys or HDL-C <50 mg/dL for girls, and
  * non-HDL-C ≥120 mg/dL
* Participant consent, or parental/guardian consent and participant assent

Exclusion Criteria:

* Current use of lipid lowering medication, growth hormone, systemic corticosteroids, cyclosporine, protease inhibitors, erythromycin, rifampin, colchicine, warfarin, second generation psychotropic drugs, oral isotretinoin; stable doses of stimulant or antidepressant therapy and antihypertensive medications will be accepted
* Known allergy or hypersensitivity to statin
* Patients who have had bariatric surgery or plan to have bariatric surgery during the trial
* Female who is pregnant, plans to become pregnant or is sexually active without contraception
* Uncontrolled stage 2 hypertension (systolic or diastolic blood pressure ≥95th percentile for age, sex and height percentile + 12 mmHg or ≥140/90, whichever is lower for participants <13 years of age; ≥140/90 for participants ≥13 years of age) confirmed after an appropriate evaluation
* Diabetes (type 1 or type 2) by American Diabetes Association criteria (fasting glucose ≥126 mg/dL, HbA1c ≥6.5%, random glucose ≥200 mg/dL, or 2-hour oral glucose tolerance testing glucose ≥200 mg/dL)
* Use of insulin sensitizing therapy
* Known renal insufficiency (known chronic renal disease, estimated glomerular filtration rate (GFR) <60 mL/min/1.73m2 at screening)
* Uncontrolled thyroid disease (TSH at screening >1.5x upper limit of normal, clinical or other laboratory evidence of hypothyroidism, or thyroid hormone therapy that has not been stable for 6 weeks prior to screening)
* Proteinuria suggestive of renal disease (more than trace together with an elevated urine protein:creatinine ratio as per local lab)
* Syndromic patients or patients with neurocognitive delay precluding adherence with study drug
* Liver disease other than non-alcoholic fatty liver disease (NAFLD) either diagnosed or suggested by alanine aminotransferase (ALT) ≥ 40 U/L, or severe NAFLD indicated by ALT ≥ 200 U/L
* Unexplained persistent elevated creatine kinase (CK) level >3x upper limit of normal
* Plans to leave the geographic area before completion of the anticipated 2 years of trial participation
* Any unstable medical or emotional condition or chronic disease that would preclude following the protocol or impact valid vascular measurement
* Admits to current smoking, current alcohol consumption

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
the effect of pitavastatin versus placebo on vascular measures in at least 354 obese adolescents with combined dyslipidemia of obesity (CDO) | 2 years
  Pulse wave velocity (PWV)

SECONDARY OUTCOMES:
the effect of pitavastatin versus placebo on vascular measures in obese adolescents with combined dyslipidemia of obesity (CDO) | 2 years
  carotid intima media thickness (CIMT)
the effect of pitavastatin versus placebo on vascular measures in at least 354 obese adolescents with combined dyslipidemia of obesity | 2 years
  carotid artery stiffness
the effect of pitavastatin versus placebo on Standard Fasting Lipid Profile (FLP) | 2 years
  Change in time in standard fasting lipid profile
the effect of pitavastatin versus placebo on lipid measures | 2 years
  Change in time in apolipoproteins
the effect of pitavastatin versus placebo on Nuclear magnetic resonance (NMR) Spectroscopy Lipoprotein Particle Assessment | 2 years
  Change in time in NMR Spectroscopy Lipoprotein Particle Assessment
the effect of pitavastatin versus placebo on composite outcome of Number of Participants With Abnormal Laboratory Values and/or Adverse Events | 2 years
  Number of abnormal (yes/no) lab values based on Liver function tests (ALT, AST); creatine kinase (CK), muscle symptoms; markers of glycemic control/development of diabetes (fasting plasma glucose, HgbA1c) and change in surrogate markers of insulin sensitivity (fasting insulin, C-peptide, Homeostatic model assessment Insulin resistance (HOMA-IR), 1/insulin, QUICKI); height velocity (change in height z score) and adverse events
the effect of pitavastatin versus placebo on prevalence of adverse events. | 2 years
  Number of adverse events and other subject-reported symptoms (including neurocognitive and depressive symptoms).
the effect of pitavastatin versus placebo on prevalence of abnormal Liver function tests (ALT, AST) | 2 years
  Number of abnormal (yes/no) lab values based on Liver function tests (ALT, AST)
the effect of pitavastatin versus placebo on prevalence of abnormal creatinine kinase (CK) tests | 2 years
  Number of abnormal (yes/no) lab values based on creatinine kinase (CK) tests
the effect of pitavastatin versus placebo on composite outcome of markers of glycemic control/development of diabetes | 2 years
  Number of abnormal (yes/no) lab values based on markers of glycemic control/development of diabetes (fasting plasma glucose, HgbA1c)
the effect of pitavastatin versus placebo on composite outcome of abnormal change in surrogate markers of insulin sensitivity | 2 years
  Number of abnormal (yes/no) lab values based on change in surrogate markers of insulin sensitivity (fasting insulin, C-peptide, HOMA-IR)
the effect of pitavastatin versus placebo on prevalence of abnormal changes in height | 2 years
  Number of abnormal (yes/no) values based on change in height in time

CONTACTS AND LOCATIONS:
Locations (16):
- United States (15):
  - Nemours/Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] de Ferranti SD, Teng JE, Arslanian SA, Atz AM, Brothers JA, Cartoski MJ, Freemon DR, Magge SN, Mahle WT, Mietus-Snyder M, Peterson A, Raghuveer G, Russell MW, Shah AS, Sponseller CA, Stylianou M, Trachtenberg FL, Urbina EM, Ware AL, Zachariah J, Zadokar VV, McCrindle BW; Pediatric Heart Network Investigators. A multicenter trial to test pitavastatin calcium in youth with combined dyslipidemia of obesity: Design, implementation, challenges, and responses. Am Heart J. 2025 Dec 15;294:107327. doi: 10.1016/j.ahj.2025.107327. Online ahead of print. PMID 41407061